CLINICAL TRIAL: NCT01255683
Title: Single-arm Clinical Evaluation of Oral Steroid Treatment for Chronic Rhinosinusitis
Brief Title: Oral Steroid Treatment for Chronic Rhinosinusitis
Status: Withdrawn | Type: Observational
Why Stopped: Lack of proposed funding.
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Timothy L. Smith, MD, MPH, Oregon Health & Science University
Other Study IDs: unfunded2
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2010-12

CONDITIONS: Chronic Rhinosinusitis
Keywords: Chronic; Sinusitis; Steroid; treatment
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Sinusitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic rhinosinusitis
  Interventions: Drug: oral corticosteroid taper

INTERVENTIONS:
Drug: oral corticosteroid taper — This is an observational study in which patients self-select oral steroid treatment for symptoms of CRS. Drug treatments are NOT assigned in this investigation.

SUMMARY:
Despite the common use of oral steroids in the management of chronic rhinosinusitis (CRS), the natural history and efficacy of this treatment modality has not been fully elucidated. Specifically, patients who have undergone prior ESS and have recalcitrant CRS, the natural history of endoscopic improvement and quality of life (QoL) outcomes, following an oral steroid taper, is poorly defined. The purpose of this non-randomized single-arm clinical trial is to evaluate the effectiveness of an oral steroid taper in improving endoscopic grading, QoL, and olfactory function as well as defining the duration of improvement, in patients with recalcitrant CRS with prior endoscopic sinus surgery (ESS).

ELIGIBILITY:
Inclusion Criteria:

* Adult ( > 18 years of age)
* CRS defined by 2007 Adult Sinusitis Guidelines.12
* Subject must be able to complete QoL questionnaires written in English
* Previous sinus surgery including unilateral or bilateral total ethmoidectomy
* Minimum nasal blockage score on SinoNasal Outcomes Test-22 (SNOT-22) > 3
* Severe sinonasal inflammation where the next treatment option is a 12- day oral prednisone taper
* Obstruction of the ethmoid sinus region or middle meatus eligible for revision endoscopic sinus surgery
* Lund-Kennedy endoscopy score > 4
* Elects 12-day tapering dose of oral steroids (Prednisone) as a next treatment option

Exclusion Criteria:

* Unable to complete questionnaires or clinical testing or cooperate with study evaluations in English
* Contra-indication to oral steroids
* Endoscopic sinus surgery < 3 months of presentation
* Completed course of oral corticosteroids within the previous 3 month period
* Subjects presenting with unilateral chronic rhinosinusitis
* Pregnancy or possibility to become pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult study population with a confirmed diagnosis of chronic sinusitis presenting to the tertiary rhinology clinic at Oregon Health & Science University (OHSU).
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-12; Primary Completion 2011-11 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Health-related quality-of-life | Change from baseline to 6 months
  The two main outcome measures to evaluate changes in QoL include the Sinonasal Outcome Test-22 (SNOT-22) and Nasal Obstruction Scoring Evaluation (NOSE) instruments. The SNOT-22 is a validated, 22-item outcome measure applicable to both sinonasal conditions and surgical treatments (score range: 0-110). Lower total scores on the SNOT-22 imply better QoL. The SNOT-22 will be administered by the Study Coordinator to study participants at baseline, as well as 2 week, 1 month, 3 month, and 6 month follow-up appointments.

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States